CLINICAL TRIAL: NCT03242616
Title: Randomized Phase II Trial of Pemetrexed Plus Vinorelbine Versus Vinorelbine in Patients With Recurrent or Metastatic Breast Cancer Previously Treated With or Resistant to Anthracycline and Taxane
Brief Title: PemVin vs Vin in Previously Treated Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H1607-172-780
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pemetrexed + Vinorelbine (Experimental): Vinorelbine (25 mg/m2, day 1 & 8)
  * Pemetrexed (500 mg/m2, day 1)
    1. Actinamide 1mg IM: 1 week before 1st dose, q 9 weeks (1wk before 1st cycle, 4th,7th,10th…. cycle after then.)
    2. Folic acid 1mg daily: 1 week before 1st dose until 3 weeks after last dose
    3. Dexa 4mg po bid on D0-2
  Interventions: Drug: Pemetrexed + Vinorelbine
- Vinorelbine (Active Comparator): Vinorelbine (25 mg/m2, day 1 & 8)
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Pemetrexed + Vinorelbine — Vinorelbine (25 mg/m2, day 1 & 8)
  * Pemetrexed (500 mg/m2, day 1)
  Arms: Pemetrexed + Vinorelbine
Drug: Vinorelbine — Vinorelbine (25 mg/m2, day 1 & 8)
  Arms: Vinorelbine

SUMMARY:
Pemetrexed is a multi-targeted anti-folate, that is used for non-small cell lung cancer and mesothelioma. There are several clinical studies of pemetrexed in breast cancer, but these are largely done before the wide use of premedication (steroid and vitamin B12) for pemetrexed. Moreover, it has not been studied in combination with vinorelbine, which is a commonly used drug for anthracycline- and taxane-pretreated metastatic breast cancer.

This is a randomized phase II study of pemetrexed plus vinorelbine versus vinorelbine in patients with recurrent or metastatic breast cancer previously treated with or resistant to an anthracycline and taxane.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed, recurrent or metastatic breast cancer
2. HER2-negative
3. ECOG PS 0-2
4. Age ≥ 20 years
5. Anthracycline- and Taxane-pretreated
6. Wash-out period of 3 weeks for cytotoxic chemotherapy
7. Wash-out period of 2 weeks for hormone therapy or radiotherapy
8. measurable or non-measurable lesions by RECIST v1.1
9. Adequate hematological functions : ANC ≥1,500/mm3, Platelet ≥100,000/mm3, Hb≥ 9g/dL
10. Adequate liver functions
11. Adequate renal functions : sCr≤1.5mg/dL
12. Subjects willing to follow study protocol
13. Informed consent before study entry

Exclusion Criteria:

1. More than 3 lines of chemotherapy for metastatic breast cancer
2. Pregnant or breastfeeding women
3. Previous exposure to Pemetrexed or Vinorelbine
4. Neuropathy (grade 2 or more)
5. Symptomatic CNS metastasis
6. History of malignant disease within 5 years (except for cured basal cell cancer or squamous cell cancer of skin, cured thyroid cancer, in-situ cervical cancer)
7. Hypersensitivity to study medication or related drugs
8. Concomitant vaccination for yellow fever

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
progression free survival | response assessment every 6 weeks, for up to 2 years
  From date of first dose of study drug till the date of documented progression or death from any cause

SECONDARY OUTCOMES:
response rate | response assessment every 6 weeks, for up to 2 years
  Proportion of patients with objective response by RECIST version 1.1
duration of response | response assessment every 6 weeks, for up to 2 years
  Time from documentation of tumor response to disease progression
overall survival | up to 2 years
  From date of first dose of study drug till the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No